CLINICAL TRIAL: NCT00978289
Title: Microenvironment of Adipose Tissue in Endocannabinoid System Before and After Roux-en-y Gastric Bypass Surgery
Brief Title: Microenvironment of Adipose Tissue in Endocannabinoid System
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Naji Abumrad, Chairman, Department of Surgery, Vanderbilt University
Other Study IDs: IRB#080516
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Obesity
Keywords: obesity; gastric bypass surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, adipose tissue, adipose tissue microdialysate
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is examine the relationship between adipose tissue inflammation and activation of the endocannabinoid system before and after Roux-en-Y gastric bypass surgery. The investigators hypothesize that the metabolic improvements and weight loss are due to mechanisms that antagonize the endocannabinoid system.

ELIGIBILITY:
Inclusion Criteria:

* BMI>35 kg/m2
* Age 20-60 yrs
* Approved and scheduled for gastric bypass surgery
* Stable body weight for past 3 months

Exclusion Criteria:

* Positive pregnancy test
* Previous gastric surgeries
* Intercurrent infections
* History of ketoacidosis or current metabolic acidosis
* Serum creatinine or liver function tests > 2 times upper limits of normal
* Taking drugs that are known to affect carbohydrate or lipid metabolism other than anti-diabetes mediations.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects approved and scheduled for gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naji Abumrad, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States